CLINICAL TRIAL: NCT00003075
Title: A Randomized Double-Blind Study of N-(4-hydroxyphenyl) Retinamide (4-HPR) Versus Placebo in Patients With Cervical Intraepithelial Neoplasia (CIN) Grade 2-3
Brief Title: Fenretinide in Treating Patients With Cervical Neoplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ID92-027; P30CA016672 (NIH); MDA-ID-92027 (Other: UT MD Anderson Cancer Center); NCI-P97-0092; CDR0000065761 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-05-27 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenretinide (Experimental)
  Interventions: Drug: Fenretinide
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenretinide — Oral Fenretinide daily for 6 months with 3 days of rest every month.
  Other Names: 4-HPR
  Arms: Fenretinide
Other: Placebo — Oral placebo daily for 6 months with 3 days of rest every month.
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention uses drugs to try and prevent development of cancer. Fenretinide may be effective in treating cervical neoplasia and preventing cervical cancer.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of fenretinide to placebo in treating patients with cervical neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of fenretinide (N-(4-hydroxyphenyl) retinamide; 4-HPR) at regressing cervical intraepithelial neoplasia (CIN). II. Document the qualitative and quantitative toxicity of 4-HPR in women with CIN.

OUTLINE: This is a double blinded study. Patients are randomized to receive either fenretinide or placebo. Patients are administered fenretinide or a placebo by mouth (PO) daily for 6 months with 3 days of rest every month. Patients undergo colposcopy, colpophotography, and Pap smears at 3, 6, 9, and 12 months. Patients undergo cervical biopsy at 6 and 12 months to assess changes.

PROJECTED ACCRUAL: 84-100 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed new or recurrent cervical intraepithelial neoplasia grade 2-3 lesion involving at least one quadrant of the transformation zone of the cervix

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 months Hematopoietic: Absolute granulocyte count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Other: Fertile patients must use effective contraception Fasting triglyceride less than 2 times normal No prior malignancy Must consent to colposcopy and cervical biopsy

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1993-03-05 (Actual); Primary Completion 2001-05-01 (Actual); Study Completion 2001-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Fenretinide at Regressing CIN | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org